CLINICAL TRIAL: NCT00970203
Title: Feasibility, Safety and Efficacy Evaluation of Alpha-Type 1 Dendritic Cell(DC)-Based Vaccines Loaded With Allogeneic Prostate Cell Lines in Combination With Androgen Ablation in Patients With PSA Progression After Local Therapy for Prostate Cancer
Brief Title: Dendritic Cell (DC)-Based Vaccines Loaded With Allogeneic Prostate Cell Lines in Combination With Androgen Ablation in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06-070
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2020-05-07 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Cancer of Prostate; Cancer of the Prostate; Neoplasms, Prostate; Neoplasms, Prostatic; Prostate Cancer; Prostate Neoplasms; Prostatic Cancer
Keywords: Vaccine; Androgen Ablation; PSA Progression
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A (Experimental): 3 months of androgen ablation followed at PSA progression by 3 months of the combination of androgen ablation + DC1 vaccine
  AA: Lupron 22.5 mg or Zoladex 10.8 mg DC vaccine: intradermal (id) vaccine of 3-5 x 10e6 cells
  Interventions: Biological: androgen ablation (AA); Biological: DC1 vaccine
- Cohort B (Experimental): 3 months of the combination of androgen ablation + DC1 vaccine followed at PSA progression by 3 months of androgen ablation
  AA: Lupron 22.5 mg or Zoladex 10.8 mg DC vaccine: intradermal (id) vaccine of 3-5 x 10e6 cells
  Interventions: Biological: androgen ablation (AA); Biological: DC1 vaccine

INTERVENTIONS:
Biological: androgen ablation (AA) — Lupron 22.5 mg or Zoladex 10.8 mg
Biological: DC1 vaccine — 3-5 x 10e6 cells total
  Other Names: alpha dendritic cell 1 vaccine

SUMMARY:
This study will evaluate the feasibility, safety, and efficacy of intradermal vaccination of prostate cancer patients with alpha-type-1-polarized dendritic cells (DC1) loaded with apoptotic allogeneic tumor (LNCap). The study will target men with recurrent prostate cancer, who failed local therapy, have no measurable metastasis, but have a rising PSA with a doubling time of less than 10 months. The selection of this study group enables us to evaluate time to PSA progression, a highly relevant, clinical primary endpoint of efficacy in this two arm study. In order to facilitate infiltration of vaccination-induced T cells into tumor site(s) and to reduce tumor-specific tolerance, subjects will receive the vaccine in combination with limited androgen ablation (AA) with a LHRH analogue for 3 months. Subjects will be randomly assigned to one of two cohorts. In cohort A subjects will be first treated with limited AA alone for 3 months, and at the time of PSA relapse (PSA ≥ 1 ng/dL) will receive the DC vaccine in conjunction with AA. In cohort B, the sequence of treatment will be reversed. Efficacy will be estimated as the within-subject difference in time to PSA relapse following the combination treatment as compared to the AA alone, thus, each subject will serve as his own control. All subjects will commence the DC1-based vaccination 2 weeks prior to treatment with the LHRH analogue. Each subject will receive 1 intradermal (i.d.) dose of the vaccine at weeks 1, 5, 9, and 13 for a total of 4 doses. Additional courses of vaccination may be administered to subjects without evidence of disease progression every 3 months (±1 month) for up to 12 months depending on the number of doses originally produced and available after the 4 intended protocol doses. All doses of the vaccine will be administered intradermally (i.d.).

DETAILED DESCRIPTION:
Dendritic cells or "DCs" are special white blood cells that stimulate the immune system. This study is being done to test the feasibility, safety and efficacy of a specific type of dendritic cell when injected under the skin of patients with prostate cancer. The researchers conducting this study will evaluate the time to prostate specific antigen (PSA) progression and will also be performing tests to see how the immune system is responding to the injections.

This is a 2 group crossover trial in which patients are randomly assigned to one of two treatment arms:

A. 3 months of androgen ablation (AA) to be followed at PSA progression by 3 months of the combination of AA and alpha-type 1 dendritic cell vaccine (DC1); B. 3 months of the combination of AA and alpha-type 1 dendritic cell vaccine followed at PSA progression by 3 months of AA.

Primary Objectives

* Feasibility objective: the ability to successfully generate and administer the alpha-DC1 vaccine.
* Safety objective: assess the tolerability and toxicity of the alpha-DC1 vaccine.
* Efficacy objective: evaluate the effect of the alpha-DC1 vaccine on time to PSA progression compared to AA alone. PSA progression is defined as a rise in the PSA value to e 1.0 ng/mL.

Secondary Objectives

* To determine the change in PSA velocity prior to and following the proposed treatment.
* To evaluate (in all subjects) the vaccination-induced DTH responses to LNCap, the cell line vaccine, and to compare this with vaccination-induced responses to tumor-untreated antigen (KLH).
* To evaluate the vaccination-induced changes of Th1/Th2 profiles of the responses to PAP and PSMA.
* To evaluate the CTL responses in blood to the whole LNCap cells (in all subjects) and (in all subjects who are HLA-A2 positive) the CTL responses to HLA-A2.1 restricted peptides derived from PAP and PSMA.
* To comprehensively evaluate the CD4+ and CD8+ T cell responses (fine specificity and Th1/Th2/Treg cytokine profile) to the previously-identified and novel immunogenic epitopes of PAP and PSMA, using the EPIMAX system.

This is a 2 group crossover trial in which patients are randomly assigned to one of two treatment arms:

A. 3 months of androgen ablation (AA) to be followed at PSA progression by 3 months of the combination of AA and alpha-type 1 dendritic cell vaccine (DC1); B. 3 months of the combination of AA and alpha-type 1 dendritic cell vaccine followed at PSA progression by 3 months of AA.

In this crossover trial each patient will serve as their own control. Following either therapy the time to PSA progression, defined as the time between treatment and the first instance of PSA increase to 1ng/ml. The endpoint is the difference between time to PSA progression for the combination of AA + DC1 compared to AA alone. A total of 12 evaluable patients (6 patients/arm) will be enrolled on the trial. Patients who do not complete both courses (AA and AA+DCV) will be replaced. This schema will also help us better estimate the time to PSA recovery following 3 months of limited androgen ablation in our cohort of patients.

All patients in Cohort B, will commence DC1-based vaccination 2 weeks prior to treatment with the LHRH analogue. Each patient will receive four i.d. doses of the vaccine at weeks 1, 4, 8, and 12. The LHRH analogue (Lupron 22.5 mg or Zoladex 10.8 mg), will be administered 2 weeks after the 1st dose of the DC vaccine. Additional courses of vaccination can be administered to any patients without evidence of disease progression, every 3 months for up to 12 months.

Patients will undergo a thorough pre-study evaluation, and then undergo leukapheresis to generate the DC-based vaccine. Each patient will receive 4 doses of intradermal (i.d.) DC1-based vaccine at weeks 1, 4, 8, and 12.

ELIGIBILITY:
Eligibility Criteria

* Patients with histologically proven prostate cancer and tumors limited to the prostate (including seminal vesicle involvement, provided all visible disease was surgically removed) who have completed local therapy and have an elevated PSA after surgery or rising PSA after radiation therapy, as defined below.
* Age 18 years or older
* Histologically confirmed diagnosis of prostate cancer.
* Previous treatment with definitive surgery or radiation therapy or both.
* No evidence of metastatic disease on physical exam, CT/MRI/CXR (see Section 7.1 for radiologic imaging), and bone scan within 4 weeks prior to randomization.
* Prior neoadjuvant/adjuvant hormonal, androgen deprivation therapy, or chemotherapy is allowed if it was last used > 12 months prior to first vaccination.
* No therapy modulating testosterone levels (such as leuteinizing-hormone releasing-hormone agonists/antagonists and antiandrogens) is permitted within 12 months prior to first vaccination. Agents such as 5α-reductase inhibitors, ketoconazole, megestrol acetate, systemic steroids (replacement doses of steroids are allowed), PC-SPES, and Saw Palmetto are not permitted at any time during the period that the PSA values are being collected.
* Hormone-sensitive prostate cancer as evident by a serum total testosterone level > 150 ng/dL or > 6 nmol/L at the time of enrollment within 4 weeks prior to randomization.
* All patients must have evidence of biochemical progression as determined by a reference PSA value followed by 1 confirmatory rising PSA value, higher than the previous value, obtained at least 2 weeks apart. All of these PSA values must be obtained at the same reference lab, and all must be done within 6 months prior to enrollment.
* The most recent of the PSA values must be ≥ 2.0 ng/mL. This measurement must be obtained within 1 month prior to enrollment.
* The PSA doubling time (PSA-DT) must be less than 12 months.
* ECOG performance status 0 or 1.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count > 1,500/µL
  * Platelets > 100,000/µL
  * Total bilirubin 1.5 x upper limit of normal (ULN)
  * SGOT (AST) and SGPT (ALT) < 2.5 x institutional ULN
  * Creatinine 1.5 x ULN
* The effects of dendritic cell vaccines on the developing human fetus are unknown. For this reason men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.

Exclusion Criteria

* Patients must not be receiving other investigational agents or concurrent anticancer therapy.
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not have active eczema, atopic dermatitis, or other exfoliative skin conditions (e.g., burns, impetigo, varicella zoster, severe acne, contact dermatitis, psoriasis, herpes or other open rashes or wounds).
* Presence of an active acute or chronic infection, including urinary tract infection, HIV or viral hepatitis. HIV patients are excluded based on immunosuppression which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections. If clinically indicate, HIV/viral hepatitis testing will be performed to confirm status.
* Patients with a history of auto-immune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Patients receiving replacement thyroid hormone would be eligible.
* No concurrent use of systemic steroids, except for local (topical, nasal, or inhaled) steroid use. Adrenal replacement doses of corticosteroids are allowed.
* Subjects with concurrent additional malignancy (with exception of non-melanoma skin cancers and superficial bladder cancer or malignancy within last 3 years).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2018-10-05 (Actual); Study Completion 2019-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard J Appleman, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer institute, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: 3 months of androgen ablation followed at PSA progression by 3 months of the combination of androgen ablation + DC1 vaccine
  AA: Lupron 22.5 mg or Zoladex 10.8 mg DC vaccine: intradermal (id) vaccine of 3-5 x 10e6 cells
  androgen ablation (AA): Lupron 22.5 mg or Zoladex 10.8 mg
  DC1 vaccine: 3-5 x 10e6 cells total
- Cohort B: 3 months of the combination of androgen ablation + DC1 vaccine followed at PSA progression by 3 months of androgen ablation
  AA: Lupron 22.5 mg or Zoladex 10.8 mg DC vaccine: intradermal (id) vaccine of 3-5 x 10e6 cells
  androgen ablation (AA): Lupron 22.5 mg or Zoladex 10.8 mg
  DC1 vaccine: 3-5 x 10e6 cells total
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (6.9) | 64 (6.4) | 64 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients to Successfully Generate and Administer the Alpha-DC1 Vaccine
Description: The percentage of patients for which the alpha-DC1 vaccine was generated and for which 4 vaccine injections were administered (1 injection every 4 weeks).
Time Frame: 16 weeks
Population: All treated and eligible patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 7 | 6
percentage of participants | 100 [70.1 to 100] | 100 [67. to 100]

2. Primary Outcome: Tolerability and Toxicity of the Alpha-DC1 Vaccine
Description: The percentage of patients who experienced vaccine related toxicity.
Time Frame: 16 weeks
Population: All treated and eligible patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 7 | 6
percentage of participants | 0 [0 to 29.2] | 0 [0 to 33]

3. Primary Outcome: The Effect of the DC1 Vaccine on Time to PSA Progression Compared to AA Alone
Description: The mean difference between time to relapse on androgen ablation plus alpha DC-1 vaccine vs androgen ablation
Time Frame: Approximately 18 months
Population: Despite numerous attempts to obtain required data from the previous IND holder where the data is housed, including attempts to contact study PI and team, no responses were obtained and no data are available for this Outcome Measure.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in PSA Velocity Prior to and Following the Proposed Treatment.
Time Frame: Approximately 18 months
Population: The IND holder where the data is housed has stated that the data for this outcome was not collected.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Evaluate (in All Subjects) the Vaccination-induced DTH Responses to LNCap, the Cell Line Vaccine, and to Compare This With Vaccination-induced Responses to Tumor-untreated Antigen (KLH)
Time Frame: Approximately 17 weeks
Population: The IND holder where the data is housed has stated that the data for this outcome was not collected.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Evaluate the Vaccination-induced Changes of Th1/Th2 Profiles of the Responses to PAP and PSMA
Time Frame: Approximately 18 to 24 months
Population: The IND holder where the data is housed has stated that the data for this outcome was not collected.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Evaluate the CTL Responses in Blood to the Whole LNCap Cells (in All Subjects) and (in All Subjects Who Are HLA-A2 Positive) the CTL Responses to HLA-A2.1 Restricted Peptides Derived From PAP and PSMA
Time Frame: Approximately 18 to 24 months
Population: The IND holder where the data is housed has stated that the data for this outcome was not collected.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Comprehensively Evaluate the CD4+ and CD8+ T Cell Responses (Fine Specificity and Th1/Th2/Treg Cytokine Profile) to the Previously-identified and Novel Immunogenic Epitopes of PAP and PSMA, Using the EPIMAX System
Time Frame: Approximately 18 to 24 months
Population: The IND holder where the data is housed has stated that the data for this outcome was not collected.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Between 6 and 18 months.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=7) | Cohort B (N=6)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Scleral disorder (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Edema trunk (General disorders) | 0 | 1
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 4
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 3
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Hot flashes (Vascular disorders) | 6 | 6
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Despite numerous attempts to obtain required data from the previous IND holder where the data is housed, including attempts to contact study PI and team, no responses were obtained and no data were available for this some Outcome Measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT00970203/Prot_SAP_000.pdf